CLINICAL TRIAL: NCT02202031
Title: Controlling Urgency Through Relaxation Exercises
Acronym: CURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Alison Huang, MD, Assistant Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-13319; 1R01AG047894 (NIH)
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Overactive Bladder; Urgency Urinary Symptoms; Urgency Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Music Therapy (Experimental): Participants will use an identical appearing device, programmed to play quiet, relaxing music, while monitoring spontaneous breathing. Participants will be instructed to use their devices for at least 15 minutes per day for 12 weeks.
  Interventions: Behavioral: Music Therapy
- Paced Respiration (Experimental): Participants will use a small, commercially-available guided-breathing device to practice breathing at a rate slower than 10 breaths per minute. Participants will be instructed to use their devices for at least 15 minutes per day for 12 weeks.
  Interventions: Behavioral: Paced Respiration

INTERVENTIONS:
Behavioral: Paced Respiration — Participants will use a small, commercially-available guided-breathing device to practice breathing at a rate slower than 10 breaths per minute. Participants will be instructed to use their devices for at least 15 minutes per day for 12 weeks.
  Arms: Paced Respiration
Behavioral: Music Therapy — Participants will use an identical appearing device, programmed to play quiet, relaxing music, while monitoring spontaneous breathing. Participants will be instructed to use their devices for at least 15 minutes per day for 12 weeks.
  Arms: Music Therapy

SUMMARY:
We propose to conduct a rigorous, 12-week, randomized controlled trial of two relaxation therapies in 160 ambulatory women who report an average of at least 3 urgency-associated voiding or incontinence episodes per day. Participants will be randomized in a 1:1 ratio to: 1) practice slowing their resting respiratory rate to 5 to 10 breaths per minute for at least 15 minutes/day at home using a portable guided-breathing device; or 2) use an identical-appearing device that plays relaxing music while monitoring their spontaneous breathing pattern. We do not know if either of the two types of relaxation therapies is effective in treating OAB. All women will also receive a usual care pamphlet providing basic information about other traditional self-management strategies for OAB.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 21 years or older who are able to walk to the bathroom without assistance
2. Report recurrent episodes of urgency (sudden or strong urges to urinate) beginning at least 3 months prior to screening
3. Able to record all voiding and incontinence episodes on a screening 3-day voiding diary29,30 and rate the severity of urgency associated with each episode using a validated urgency severity scale31
4. Document at least 9 voiding or incontinence episodes on the above 3-day voiding diary that are associated with at least moderate sensation of urgency (using the above validated urgency severity scale) 31
5. Willing to refrain from initiating other treatments that may affect voiding pattern during the trial period

Exclusion Criteria:

1. Use of anticholinergic OAB medications or other medications known to affect urinary function (i.e., diuretics, tricyclic antidepressants) within 1 month of screening
2. Current urinary tract infection (detected via screening dipstick urinalysis or urine culture) or a history more than 3 urinary tract infections in the preceding 1 year
3. Prior history of lower urinary tract surgery, pelvic cancer, or pelvic irradiation; or other pelvic or abdominal surgery within 6 months of screening
4. History of interstitial cystitis, fistula in the bladder or rectum, or congenital or childhood defect leading to chronic urinary incontinence, retention, or other chronic urinary symptoms
5. Known history of major neurologic conditions likely to have major or permanent effects on bladder function such as stroke, multiple sclerosis, spinal cord injury, or Parkinson's disease
6. Use of bladder botulinum injections, electrostimulation, or other invasive therapies for OAB or incontinence within 3 months of screening
7. Formal pelvic floor rehabilitation or other formal behavioral therapy for bladder symptoms involving a physical therapist or other certified practitioner within 3 months of screening
8. Started, stopped, or changed dosage of a psychoactive medication likely to affect anxiety (SSRIs/SNRIs, tricyclics) within 3 months of screening, or plans to start, stop, or change dosage during the trial
9. Resting blood pressure (average of 2 measures) less than 100/60 at screening (women with baseline low blood pressure may theoretically be at increased risk of hypotension with use of RESPeRATE)
10. Resting breathing rate already below 10 breaths/minute before treatment (as measured during run-in)
11. History of chronic pulmonary disease likely to interfere with breathing exercises (e.g., emphysema)
12. Currently pregnant, gave birth within the past 3 months, or planning pregnancy during the study period
13. Unable or willing to sign an informed consent, fill out questionnaires, or undergo study procedures

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Huang, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Music Therapy: Participants will use an identical appearing device, programmed to play quiet, relaxing music, while monitoring spontaneous breathing. Participants will be instructed to use their devices for at least 15 minutes per day for 12 weeks.
  Music Therapy
- Paced Respiration: Participants will use a small, commercially-available guided-breathing device to practice breathing at a rate slower than 10 breaths per minute. Participants will be instructed to use their devices for at least 15 minutes per day for 12 weeks.
  Paced Respiration
Period: Overall Study
Arm/Group | Music Therapy | Paced Respiration
Started | 82 | 79
Completed | 77 | 74
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Too Busy | 1 | 3
Not completed — Illness/Medical Reason | 0 | 2
Not completed — Intolerance/Lack of Improvement | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Music Therapy | Paced Respiration | Total
Number analyzed (Participants) | 82 | 79 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.67 (10.9) | 60.35 (11.4) | 61.02 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 79 | 161
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Asian-American | 6 | 7 | 13
  Latina | 6 | 12 | 18
  Mixed | 7 | 3 | 10
  Non-Latina African-American | 12 | 12 | 24
  Non-Latina White | 49 | 40 | 89
  Unknown | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 82 | 79 | 161
Incontinence Frequency [Mean (Standard Deviation); unit: Episodes per day] — Measure Description: Urge incontinence is a sudden and strong need to urinate. Urinary incontinence is the involuntary leakage of urine.
  Episodes per day
    Urgency Incontinence | 1.19 (1.6) | 1.37 (2.0) | 1.28 (1.8)
    Moderate Sensation of Urgency Incontinence or Void | 6.77 (3.8) | 7.10 (2.9) | 6.93 (3.4)
    Severe Sensation of Urgency Incontinence or Void | 2.42 (2.3) | 3.01 (2.6) | 2.71 (2.4)
    Daytime voiding | 9.70 (3.8) | 9.81 (2.8) | 9.76 (3.3)
    Nighttime voiding | 1.42 (1.0) | 1.25 (1.0) | 1.34 (1.0)
    Total voiding | 11.12 (3.9) | 11.06 (2.9) | 11.09 (3.4)
Overactive Bladder Questionnaire [Mean (Standard Deviation); unit: score on a scale] — A 33-item measure of the bothersomness and impact of multiple OAB symptoms (such as urgency, incontinence, nocturia) along a 100-point scale. Higher the score the greater the bothersome.
  score on a scale | 27.59 (11.4) | 29.12 (9.9) | 28.35 (10.7)
Urgency Severity and Impact Questionnaire [Mean (Standard Deviation); unit: score on scale] — A 13-item measure of the severity and impact of urgency validated specifically in patients with Overactive Bladder (OAB). Possible score range 0-100. Higher the severity score, the more severe.
  score on scale
    Severity Subscale | 58.51 (11.7) | 58.45 (14.5) | 58.48 (13.1)
    Health-Related Quality of Life Subscale | 21.94 (15.4) | 24.57 (19.4) | 23.23 (17.5)
Urogenital Distress Inventory Short Form (UDI-6) [Mean (Standard Deviation); unit: score on scale] — A 6-item measure of the bothersomeness of multiple urinary symptoms, including urgency and incontinence. Scores range from 0-100. The higher the score, the more distress.
  score on scale | 45.19 (17.3) | 45.57 (19.6) | 45.38 (18.4)
Patient Perception of Bladder Condition (PPBC) [Mean (Standard Deviation); unit: score on scale] — A single-item assessing patient's overall perception of their bladder problems using a 6-point Likert scale. Score range of 1-6. The higher the score, the more severe.
  score on scale | 2.65 (1.0) | 2.61 (1.1) | 2.63 (1.0)
Spielberger State Trait Anxiety Inventory (STAI), Trait Component [Mean (Standard Deviation); unit: Score on scale] — A 20-item self-administered measure validated in both clinical and psychiatric populations, including patients with bladder symptoms. Scores range from 20 to 80, with higher scores indicating greater somatic anxiety.
  Score on scale | 36.82 (10.2) | 38.49 (10.5) | 37.64 (10.3)
Hospital Anxiety and Depression Scale (HADS), Anxiety Subscale [Mean (Standard Deviation); unit: score on scale] — A validated self-administered questionnaire that includes a 7-item Anxiety Subscale shown to be sensitive to change in incontinence trials.50 Scores range from 0 to 21, with higher scores indicating greater anxiety.
  score on scale | 6.22 (3.8) | 6.72 (4.0) | 6.47 (3.9)
Center for Epidemiologic Studies Depression Scale (CES-D) [Mean (Standard Deviation); unit: Score on Scale] — A 20-item measure that has been widely used in clinical trials, including trials of bladder interventions, and is sensitive to change. Total scores range from 0 to 60, with higher scores indicating greater likelihood of depression.
  Score on Scale | 10.17 (8.5) | 11.87 (10.1) | 11.01 (9.3)
Perceived Stress Scale (PSS) [Mean (Standard Deviation); unit: Score on scale] — A 10-item self-administered questionnaire assessing subjective feelings and thoughts related to perceived stress in the past month, validated in a probability sample of the United States. Scores range from 0 to 40, with higher scores indicating greater perceived stress.
  Score on scale | 13.40 (6.6) | 14.41 (7.0) | 13.89 (6.8)
Pittsburgh Sleep Quality Index (PSQI) [Mean (Standard Deviation); unit: Score on scale] — An 18-item validated questionnaire evaluating sleep quality, sleep latency, sleep efficiency, and sleep problems over a one-week period. A global sleep quality score ranging from 0 to 21 can be derived from the PSQI, with higher scores reflecting poor sleep quality.
  Score on scale | 7.11 (3.2) | 7.42 (3.8) | 7.26 (3.5)
Respiratory Sinus Arrhythmia (RSA) [Mean (Standard Deviation); unit: msec^2] — high frequency heart rate variability Population: Measure was completed by a subset of participants.
  msec^2
    Change from rest to dot task: number analyzed (Participants) | 22 | 30 | 52
    Change from rest to dot task | 0.35 (0.6) | -0.11 (0.6) | 0.08 (0.6)
    Change from rest to maze task: number analyzed (Participants) | 22 | 30 | 52
    Change from rest to maze task | -0.10 (0.6) | -0.56 (1.0) | -0.37 (0.9)
    Resting (neutral) state: number analyzed (Participants) | 22 | 30 | 52
    Resting (neutral) state | 4.75 (1.2) | 5.69 (1.6) | 5.29 (1.5)
Pre-ejection Period (PEP) [Mean (Standard Deviation); unit: msec] — The time period during which the left ventricle of the heart contracts while the aortic and mitral valves are still closed Population: Measure Analysis Population Description: Measure was completed by a subset of participants.
  msec
    Change from rest to dot task: number analyzed (Participants) | 22 | 29 | 51
    Change from rest to dot task | -3.84 (9.7) | -0.02 (6.1) | -1.67 (8.0)
    Change from rest to maze task: number analyzed (Participants) | 22 | 29 | 51
    Change from rest to maze task | -4.21 (11.6) | -0.81 (8.7) | -2.27 (10.1)
    Resting (neutral) state: number analyzed (Participants) | 22 | 29 | 51
    Resting (neutral) state | 123.07 (11.5) | 117.11 (14.8) | 119.68 (13.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Frequency of Any Voiding or Incontinence Episodes Associated With At Least a Moderate Sensation of Urgency at 12 Weeks.
Description: Self-reported on voiding diary.
Time Frame: Baseline to 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: episodes
Arm/Group | Music Therapy | Paced Respiration
Number analyzed (Participants) | 73 | 74
episodes | -1.06 [-1.74 to -0.37] | -0.86 [-1.50 to -0.13]
Statistical Analysis 1: Comparison: Music Therapy vs Paced Respiration; Test type: Superiority; p = 0.6222, ANCOVA; change from baseline, adjusted for baseline value; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.73 to 1.21]

2. Secondary Outcome: Change From Baseline in Frequency of Any Voiding or Incontinence Episodes Associated With a Severe Sensation of Urgency at 12 Weeks.
Description: Self-reported on voiding diary
Time Frame: Baseline to 12 weeks
Population: Although 77 participants randomized to Music Therapy completed week 12 visits in some form, some participants declined to complete or had missing data for one or more outcome measures at this timepoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: episodes
Arm/Group | Music Therapy | Paced Respiration
Number analyzed (Participants) | 73 | 74
episodes | -0.85 [-1.24 to -0.46] | -0.94 [-1.32 to -0.55]
Statistical Analysis 1: Comparison: Music Therapy vs Paced Respiration; Test type: Superiority; p = 0.7695, ANCOVA; change from baseline, adjusted for baseline value; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.64 to 0.47]

3. Secondary Outcome: Change From Baseline in Urgency Incontinence Episodes at 12 Weeks.
Description: Self-reported on voiding diary
Time Frame: Baseline to 12 weeks.
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: episodes
Arm/Group | Music Therapy | Paced Respiration
Number analyzed (Participants) | 73 | 74
episodes | -0.63 [-0.85 to -0.40] | -0.55 [-0.77 to -0.33]
Statistical Analysis 1: Comparison: Music Therapy vs Paced Respiration; Test type: Superiority; p = 0.6456, ANCOVA; change from baseline value, adjusted for baseline value; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.24 to 0.39]

4. Secondary Outcome: Change From Baseline in Total Voiding Episodes at 12 Weeks.
Description: Self-reported on voiding diary.
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: episodes
Arm/Group | Music Therapy | Paced Respiration
Number analyzed (Participants) | 73 | 74
episodes | -1.04 [-1.49 to -0.60] | -1.08 [-1.52 to -0.63]
Statistical Analysis 1: Comparison: Music Therapy vs Paced Respiration; Test type: Superiority; p = 0.9190, ANCOVA; change from baseline, adjusted for baseline value; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.66 to 0.60]

5. Secondary Outcome: Change From Baseline in Overactive Bladder Questionnaire Score at 12 Weeks
Description: A 33-item measure of the bothersomness and impact of multiple OAB symptoms (such as urgency, incontinence, nocturia) along a 100-point scale. Higher the score the greater the bothersome.
Time Frame: Baseline to 12 weeks.
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Music Therapy | Paced Respiration
Number analyzed (Participants) | 76 | 74
score on a scale | -15.45 [-18.03 to -12.87] | -14.29 [-16.91 to -11.68]
Statistical Analysis 1: Comparison: Music Therapy vs Paced Respiration; Test type: Superiority; p = 0.5358, ANCOVA; change from baseline, adjusted for baseline value; Mean Difference (Final Values) = 1.16, 95% CI 2-sided [-2.51 to 4.84]

6. Secondary Outcome: Change From Baseline Score of Urgency Severity and Impact Questionnaire (USIQ), Severity Subscale at 12 Weeks.
Description: A 13-item measure of the severity and impact of urgency validated specifically in patients with OAB, range of 0-100. Higher the severity score, the more severe.
Time Frame: Baseline to 12 weeks.
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Music Therapy | Paced Respiration
Number analyzed (Participants) | 76 | 74
score on a scale | -15.56 [-18.81 to -12.32] | -13.85 [-17.13 to -10.56]
Statistical Analysis 1: Comparison: Music Therapy vs Paced Respiration; Test type: Superiority; p = 0.4663, ANCOVA; change from baseline, adjusted for baseline value; Mean Difference (Final Values) = 1.72, 95% CI 2-sided [-2.90 to 6.34]

7. Secondary Outcome: Change From Baseline Score of Urgency Severity and Impact Questionnaire (USIQ), Health-Related Quality of Life Subscale at 12 Weeks.
Description: A 13-item measure of the severity and impact of urgency validated specifically in patients with OAB, range of 0-100. Higher the severity score, the more interference with quality of life.
Time Frame: Baseline to 12 weeks
Population: Although 77 participants randomized to Music Therapy and 74 participants randomized to Paced Respiration completed week 12 visits in some form, some participants declined to complete or had missing data for one or more outcome measures at this timepoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Music Therapy | Paced Respiration
Number analyzed (Participants) | 73 | 71
score on a scale | -12.35 [-15.30 to -9.39] | -10.18 [-13.17 to -7.18]
Statistical Analysis 1: Comparison: Music Therapy vs Paced Respiration; Test type: Superiority; p = 0.3134, ANCOVA; change from baseline, adjusted for baseline value; Mean Difference (Final Values) = 2.17, 95% CI 2-sided [-2.05 to 6.38]

8. Secondary Outcome: Change From Baseline in Urogenital Distress Inventory Short Form (UDI-6) Score at 12 Weeks.
Description: A 6-item measure of the bothersomeness of multiple urinary symptoms, including urgency and incontinence; scores range from 0-100. Higher the score, the more distress.
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Music Therapy | Paced Respiration
Number analyzed (Participants) | 76 | 74
score on a scale | -15.35 [-19.07 to -11.64] | -17.11 [-20.88 to -13.35]
Statistical Analysis 1: Comparison: Music Therapy vs Paced Respiration; Test type: Superiority; p = 0.5146, ANCOVA; change from baseline, adjusted for baseline value; Mean Difference (Final Values) = -1.76, 95% CI 2-sided [-7.05 to 3.53]

9. Secondary Outcome: Change From Baseline on Patient Perception of Bladder Condition (PPBC) Score at 12 Weeks.
Description: A single-item assessing patient's overall perception of their bladder problems using a 6-point Likert scale, score range 1-6. The higher the score the more severe.
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Music Therapy | Paced Respiration
Number analyzed (Participants) | 76 | 74
score on a scale | -0.74 [-0.95 to -0.53] | -0.88 [-1.09 to -0.66]
Statistical Analysis 1: Comparison: Music Therapy vs Paced Respiration; Test type: Superiority; p = 0.3611, ANCOVA; change from baseline, adjusted for baseline value; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.44 to 0.16]

10. Secondary Outcome: Change From Baseline on Spielberger State Trait Anxiety Inventory (STAI) - Trait Component Score at 12 Weeks.
Description: A 20-item self-administered measure validated in both clinical and psychiatric populations, including patients with bladder symptoms. Scores range from 20 to 80, with higher scores indicating greater somatic anxiety.
Time Frame: Baseline to 12 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Music Therapy | Paced Respiration
Number analyzed (Participants) | 76 | 74
score on a scale | -2.42 [-3.82 to -1.02] | -2.85 [-4.27 to -1.43]
Statistical Analysis 1: Comparison: Music Therapy vs Paced Respiration; Test type: Superiority; p = 0.6722, ANCOVA; change from baseline, adjusted for baseline value; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-2.43 to 1.57]

11. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) - Anxiety Subscale Score at 12 Weeks.
Description: A validated self-administered questionnaire that includes a 7-item Anxiety Subscale shown to be sensitive to change in incontinence trials. Scores range from 0 to 21, with higher scores indicating greater anxiety.
Time Frame: Baseline to 12 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Music Therapy | Paced Respiration
Number analyzed (Participants) | 76 | 74
score on a scale | -0.71 [-1.23 to -0.19] | -1.38 [-1.90 to -0.86]
Statistical Analysis 1: Comparison: Music Therapy vs Paced Respiration; Test type: Superiority; p = 0.0786, ANCOVA; change from baseline, adjusted for baseline value; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-1.4 to 0.07]

12. Secondary Outcome: Change From Baseline in Center for Epidemiologic Studies Depression Scale (CES-D) Score at 12 Weeks.
Description: A 20-item measure that has been widely used in clinical trials, including trials of bladder interventions, and is sensitive to change. Total scores range from 0 to 60, with higher scores indicating greater likelihood of depression.
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Music Therapy | Paced Respiration
Number analyzed (Participants) | 76 | 74
score on a scale | -1.97 [-3.25 to -0.69] | -3.01 [-4.31 to -1.72]
Statistical Analysis 1: Comparison: Music Therapy vs Paced Respiration; Test type: Superiority; p = 0.2284, ANCOVA; change from baseline, adjusted for baseline value; Mean Difference (Final Values) = -1.04, 95% CI 2-sided [-2.87 to 0.79]

13. Secondary Outcome: Change From Baseline in Perceived Stress Scale (PSS) Score at 12 Weeks.
Description: A 10-item self-administered questionnaire assessing subjective feelings and thoughts related to perceived stress in the past month, validated in a probability sample of the United States. Scores range from 0 to 40, with higher scores indicating greater perceived stress.
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Music Therapy | Paced Respiration
Number analyzed (Participants) | 76 | 74
score on a scale | -1.12 [-2.23 to -0.02] | -2.83 [-3.95 to -1.71]
Statistical Analysis 1: Comparison: Music Therapy vs Paced Respiration; Test type: Superiority; p = 0.0335, ANCOVA; change from baseline, adjusted for baseline value; Mean Difference (Final Values) = -1.71, 95% CI 2-sided [-3.28 to -0.13]

14. Secondary Outcome: Change From Baseline in Pittsburgh Sleep Quality Index (PSQI) Overall Sleep Quality Score at 12 Weeks.
Description: An 18-item validated questionnaire evaluating sleep quality, sleep latency, sleep efficiency, and sleep problems over a one-week period. A global sleep quality score ranging from 0 to 21 can be derived from the PSQI, with higher scores reflecting poor sleep quality.
Time Frame: Baseline to 12 weeks
Population: Although 77 participants randomized to Music Therapy and 74 participant randomized to Paced Respiration completed week 12 visits in some form, some participants declined to complete or had missing data for one or more outcome measures at this timepoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Music Therapy | Paced Respiration
Number analyzed (Participants) | 76 | 74
score on a scale | -1.22 [-1.74 to -0.70] | -1.14 [-1.67 to -0.62]
Statistical Analysis 1: Comparison: Music Therapy vs Paced Respiration; Test type: Superiority; p = 0.8408, ANCOVA; change from baseline, adjusted for baseline value; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.66 to 0.81]

15. Secondary Outcome: Change From Baseline in Respiratory Sinus Arrhythmia at 12 Weeks.
Description: Resting (neutral) state
Time Frame: Baseline to 12 weeks
Population: Although 77 participants randomized to Music Therapy and 74 participant randomized to Paced Respiration completed week 12 visits in some form, some participants declined to complete or had missing data for one or more outcome measures at this timepoint. This measure was only completed by a small subset of participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: msec^2
Arm/Group | Music Therapy | Paced Respiration
Number analyzed (Participants) | 19 | 25
msec^2 | -0.40 [-1.13 to 0.32] | -0.27 [-1.09 to 0.55]
Statistical Analysis 1: Comparison: Music Therapy vs Paced Respiration; Test type: Superiority — adjusted for baseline value, diabetes and the following medications: beta-blockers, alpha-agonists, and sympathomimetic; p = 0.5578, ANCOVA; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.32 to 0.60]

16. Secondary Outcome: Change From Baseline in Respiratory Sinus Arrhythmia (RSA) Resting (Neutral) State at 12 Weeks.
Description: Change in autonomic control as assessed by high frequency heart rate variability (RSA)
Time Frame: Baseline to 12 weeks
Population: as for outcome 15
Measure: Least Squares Mean (95% Confidence Interval); unit: msec^2
Arm/Group | Music Therapy | Paced Respiration
Number analyzed (Participants) | 19 | 25
msec^2 | -0.40 [-1.13 to 0.32] | -0.27 [-1.09 to 0.55]
Statistical Analysis 1: Comparison: Music Therapy vs Paced Respiration; Test type: Superiority; p = 0.5578, ANCOVA; Adjusted for baseline value, diabetes and the following medications: beta-blockers, alpha-agonists, and sympathomimetic

17. Secondary Outcome: Change From Baseline in Respiratory Sinus Arrhythmia (RSA) Change From Rest to Dot Task at 12 Weeks.
Description: High frequency heart rate variability
Time Frame: Baseline to 12 weeks
Population: as for outcome 15
Measure: Least Squares Mean (95% Confidence Interval); unit: msec2
Arm/Group | Music Therapy | Paced Respiration
Number analyzed (Participants) | 19 | 25
msec2 | 0.58 [-0.28 to 1.43] | 0.33 [-0.66 to 1.32]
Statistical Analysis 1: Comparison: Music Therapy vs Paced Respiration; Test type: Superiority; p = 0.7301, ANCOVA; adjusted for baseline value, diabetes and the following medications: beta-blockers, alpha-agonists, and sympathomimetic; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.79 to 0.31]

18. Secondary Outcome: Change From Baseline in Respiratory Sinus Arrhythmia (RSA) Change From Rest to Maze Task at 12 Weeks
Description: high frequency heart rate variability
Time Frame: Baseline to 12 weeks
Population: as for outcome 15
Measure: Least Squares Mean (95% Confidence Interval); unit: msec^2
Arm/Group | Music Therapy | Paced Respiration
Number analyzed (Participants) | 19 | 25
msec^2 | 0.69 [-0.09 to 1.47] | 0.26 [-0.61 to 1.13]
Statistical Analysis 1: Comparison: Music Therapy vs Paced Respiration; Test type: Superiority; p = 0.6646, ANCOVA; adjusted for baseline value, diabetes and the following medications: beta-blockers, alpha-agonists, and sympathomimetic; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-0.89 to 0.04]

19. Secondary Outcome: Change From Baseline in Pre-ejection Period (PEP) Resting (Neutral) State at 12 Weeks.
Description: PEP is the time period during which the left ventricle of the heart contracts while the aortic and mitral valves are still closed, is an established measure of sympathetic autonomic activity that can be measured non-invasively using impedance cardiography .
Time Frame: Baseline to 12 weeks
Population: as for outcome 15
Measure: Least Squares Mean (95% Confidence Interval); unit: msec
Arm/Group | Music Therapy | Paced Respiration
Number analyzed (Participants) | 18 | 24
msec | -3.41 [-21.94 to 15.12] | 0.34 [-20.19 to 20.86]
Statistical Analysis 1: Comparison: Music Therapy vs Paced Respiration; Test type: Superiority; p = 0.4993, ANCOVA; Adjusted for baseline value, diabetes and the following medications: beta-blockers, alpha-agonists, and sympathomimetic

20. Secondary Outcome: Change From Baseline in Pre-ejection Period (PEP) Change From Rest to Dot Task at 12 Weeks.
Description: The time period during which the left ventricle of the heart contracts while the aortic and mitral valves are still closed
Time Frame: Baseline to 12 weeks
Population: as for outcome 15
Measure: Least Squares Mean (95% Confidence Interval); unit: msec
Arm/Group | Music Therapy | Paced Respiration
Number analyzed (Participants) | 18 | 24
msec | 1.28 [-5.12 to 7.69] | 1.87 [-4.85 to 8.60]
Statistical Analysis 1: Comparison: Music Therapy vs Paced Respiration; Test type: Superiority; p = 0.7506, ANCOVA; adjusted for baseline value, diabetes and the following medications: beta-blockers, alpha-agonists, and sympathomimetic; Mean Difference (Final Values) = 0.59, 95% CI 2-sided [-3.05 to 4.23]

21. Secondary Outcome: Change From Baseline in Pre-ejection Period (PEP) Change From Rest to Maze Task at 12 Weeks
Description: as for outcome 20
Time Frame: Baseline to 12 weeks
Population: as for outcome 15
Measure: Least Squares Mean (95% Confidence Interval); unit: msec
Arm/Group | Music Therapy | Paced Respiration
Number analyzed (Participants) | 18 | 24
msec | -4.79 [-14.07 to 4.49] | -6.35 [-16.56 to 3.87]
Statistical Analysis 1: Comparison: Music Therapy vs Paced Respiration; Test type: Superiority; p = 0.6268, ANCOVA; adjusted for baseline value, diabetes and the following medications: beta-blockers, alpha-agonists, and sympathomimetic; Mean Difference (Final Values) = -1.55, 95% CI 2-sided [-6.98 to 3.87]

ADVERSE EVENTS:
Time Frame: Baseline to 12 weeks.
Description: At each phone and in-person contact, participants were asked about any negative changes in their health.
Arm/Group | Music Therapy | Paced Respiration
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/79
Other Adverse Events (participants affected / at risk) | 12/82 | 10/79
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Music Therapy (N=82) | Paced Respiration (N=79)
Cold/Flu (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-04): https://cdn.clinicaltrials.gov/large-docs/31/NCT02202031/Prot_SAP_000.pdf